CLINICAL TRIAL: NCT05584020
Title: Arthroscopic Anterior Cruciate Ligament Repair Versus Reconstruction for Acute Anterior Cruciate Ligament Injury: a Multicenter Randomized Controlled Surgical Trial
Brief Title: Arthroscopic Anterior Cruciate Ligament Repair Versus Reconstruction for Acute Anterior Cruciate Ligament Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0804
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL Repair (Experimental): Patients under surgical anterior cruciate ligament repair
  Interventions: Procedure: ACL Repair
- ACL Reconstruction (Other): Patients under surgical anterior cruciate ligament reconstruction
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Procedure: ACL Repair — Patients are undergoing arthroscopic anterior cruciate ligament repair. The native ACL is repaired using very strong sutures. This device is used to repair the native ACL and restore knee stability.
  Arms: ACL Repair
Procedure: ACL Reconstruction — Patients are undergoing arthroscopic anterior cruciate ligament reconstruction. The torn ligament is removed and replaced with a band of tissue that usually connects muscle to bone. The graft tendon is taken from another part of your knee or from a deceased donor.
  Arms: ACL Reconstruction

SUMMARY:
Background: Arthroscopic anterior cruciate ligament(ACL) reconstruction is so far the gold standard for the treatment of ACL ruptures, but this technique still suffers from problems of tendon-bone healing, bone tunnel enlargement, bone resorption, a low rate of return to motion,etc. In recent years, due to the innovation of medical materials and surgical techniques, anterior cruciate ligament repair technology has returned to the field of vision of clinical doctors. This technique has the advantages of preserving the natural ligaments and their proprioceptive sensation, avoiding the bone injury of the tunnel and the complications of the donor site. However, there is still a lack of high-quality clinical randomized controlled trails to provide evidence of the effect of arthroscopic ACL repair.

Hypothesis: Arthroscopic ACL repair is comparable to ACL reconstruction in patients with ACL tears (Sherman grades I and II).

Study Design: This study was a prospective, multicenter, randomized, double-blinded, parallel-controlled, non-inferiority trial design. A total of 330 patients with ACL tears were randomly divided into 2 groups, and were randomly assigned to the experimental group (arthroscopic anterior cruciate ligament repair) and the control group (arthroscopic anterior cruciate ligament reconstruction) according to 1:1. Follow-up knee function and other scores were performed at 3 months, 6 months, 1 year, and 2 years after surgery, and the total study time is expected to be 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with anterior cruciate ligament tear clearly identified by imaging or intraoperative microscope, Sherman grade I, II; planned surgery within 3 weeks after injury
2. Basic reading and writing skills, and barrier-free communication
3. A smartphone, can use WeChat or be able to learn
4. Patients give informed consent, and sign the informed consent form, and the process must meet the requirements of GCP

Exclusion Criteria:

1. Combined with other knee joint injuries (posterior cruciate ligament injury, patellar dislocation, osteoarthritis, etc.)
2. Suffering from systemic immune diseases;
3. Existing other knee joint diseases or inflammatory diseases, including osteoarthritis, cervical spine disease, rheumatoid arthritis, fibromyalgia, polymyalgia rheumatica, etc.
4. Patients who have received local hormone injection within 3 months;
5. Those who have participated in clinical trials or are undergoing other clinical trials within 3 months before screening
6. Those who have serious primary cardiovascular disease, lung disease, endocrine and metabolic disease or serious diseases that affect their survival, such as tumor or AIDS, the researchers believe that they are not suitable for selection
7. Patients with severe liver disease, kidney disease, and hematological disease, such as renal function exceeding the upper limit of the normal value, and liver function exceeding 2 times the upper limit of the normal value;
8. Suffering from viral hepatitis, infectious diseases, severe abnormal blood coagulation mechanism and other Diseases that the researchers consider inappropriate for surgery
9. Women who are pregnant or breastfeeding, or who plan to become pregnant during the follow-up period, those who have a positive urine human chorionic gonadotropin test result before sampling; menstruating women should wait until the end of menstruation before surgery;
10. Severe neurological and mental disorders Disease patients;
11. Suspected or actual history of alcohol and drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
IKDC score | 1 year
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
  Efficiency of 1 year after operation=Sum of Items/Maximum Possible Score *100

SECONDARY OUTCOMES:
IKDC score | 3 months
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items).
  Efficiency of 3 months after operation=Sum of Items/Maximum Possible Score *100
IKDC score | 6 months
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items).
  Efficiency of 6 months after operation=Sum of Items/Maximum Possible Score *100
IKDC score | 2 years
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items).
  Efficiency of 2 years after operation=Sum of Items/Maximum Possible Score *100

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China